CLINICAL TRIAL: NCT05648201
Title: Study on PhArmacokinetics of First liNe Antiretrovirals in Healthy Breastfeeding Volunteers
Acronym: PANNA-B PK
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PANNA-B PK
Record Dates: First submitted 2022-12-05; First posted 2022-12-13 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2022-12

CONDITIONS: Hiv
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — doravirine; Raltegravir Potassium; bictegravir, emtricitabine, tenofovir alafenamide, drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Doravirine (Experimental): 1 single dose of 100mg doravirine taken orally
  Interventions: Drug: Doravirine 100Mg Tab
- Raltegravir (Experimental): 1 single dose of 1200mg raltegravir taken orally
  Interventions: Drug: Raltegravir 600Mg Tab
- Biktarvy (Experimental): 1 single dose of 25/200/50mg taken orally
  Interventions: Drug: Biktarvy 50/200/25 Tab

INTERVENTIONS:
Drug: Doravirine 100Mg Tab — 1 single dose of 100mg taken orally
  Other Names: pifeltro
  Arms: Doravirine
Drug: Raltegravir 600Mg Tab — 1 single dose of 1200mg taken orally
  Other Names: issentres
  Arms: Raltegravir
Drug: Biktarvy 50/200/25 Tab — 1 single dose of 50/200/25 taken orally
  Other Names: biktarvy
  Arms: Biktarvy

SUMMARY:
No to little data exists on penetration of antiretroviral drugs in breastmilk. Too high concentrations may lead to infant toxicity and too low concentrations may lead to development of resistance in case the infant inadvertently becomes infected with the virus.

The aim of this trial is to determine the concentration of currently often used ARV (doravirine, raltegravir, bictegravir, tenofovir alafenamide, emtricitabine) in breast milk after administration of a single dose Study design: This is a single centre, single dose, open label, pharmacokinetic study in healthy volunteers.

Study population: Adult, healthy volunteers at the end of their breastfeeding period Intervention: Administration of one dose of either doravirine (DOR) 100mg, raltegravir (RAL) 1200mg or a combination of tenofovir alafenamide 25mg, emtricitabine 200mg and bictegravir 50mg (BIC/FTC/TAF).

Main study parameters/endpoints: Area under the plasma and milk concentration curve are used to calculate milk to plasma ratio.

DETAILED DESCRIPTION:
Rationale: Although current guidelines advise against breastfeeding while using antiretrovirals in people living with HIV, some women choose to breastfeed because advantages of breastfeeding may exceed the possible risk of HIV transmission to the newborn. However, no sound recommendation can be made on which antiretrovirals are most suitable during breastfeeding, because no to little data on penetration of these drugs in breastmilk exist. Too high concentrations may lead to infant toxicity and too low concentrations may lead to development of resistance in case the infant inadvertently becomes infected with the virus.

Objective: to determine the concentration of currently often used ARV (doravirine, raltegravir, bictegravir, tenofovir alafenamide, emtricitabine) in breast milk after administration of a single dose Study design: This is a single centre, single dose, open label, pharmacokinetic study in healthy volunteers.

Study population: Adult, healthy volunteers at the end of their breastfeeding period Intervention: Administration of one dose of either doravirine (DOR) 100mg, raltegravir (RAL) 1200mg or a combination of tenofovir alafenamide 25mg, emtricitabine 200mg and bictegravir 50mg (BIC/FTC/TAF).

Main study parameters/endpoints: Area under the plasma and milk concentration curve are used to calculate milk to plasma ratio.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Subjects will not directly benefit from this study, but will contribute to knowledge on breastmilk transfer of ARV and possibly enable people living with HIV to make an informed decision on breastfeeding while using these medications.

No harm is expected from participation in this study, but possible side effects should be anticipated. Known side effects of DOR are nausea (4%) and headache (3%), abnormal dreams and insomnia (1-10%), dizziness and somnolence and fatigue (1-10%). BIC/FTC/TAFs and RALs known side effects are: headache (5%), diarrhoea (5%) and nausea (4%), depression and abnormal dreams and fatigue (1-10%), suicidal ideation (0,1-1%), angio-edema (0,1-1%) and Steven Johnson syndrome (0,01-0,1%) and osteonecrosis (0,01-0,1%). Due to the fact that only one dose of the drugs will be ingested, the risk of development of one or more of these side effects is considered to be low.

Participation in this study requires subjects to be admitted for 12 hours, a visit the next morning and a return visit 7 days later. During the sampling day an intravenous indwelling catheter is installed for collection of blood samples. A total volume of 25-50ml of blood, 2 urine samples and 6 breastmilk samples (expressed using a personal electronic pump) are collected. No harm is to be expected from these sample collection procedures.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age at the moment of screening
* At least 10 days post partum
* At the end of breastfeeding period; subject is able to produce breastmilk at least two times a day and is no longer feeding infant at start of study
* Able and willing to sign an informed consent

Exclusion Criteria:

* Relevant co-medication or comorbidity that might interfere with drug absorption, distribution, metabolism or excretion
* Inability to take drugs according to the instructions (i.e. with food)
* Presence of positive HIV screening or HIV RNA
* Presence of HBsAg or HBcAg without anti-HBs
* Presence of grade III/IV anaemia (i.e. Hb <4.6 mmol/L or <7.4 g/dL).
* Presence of hereditary forms of severe galactose intolerance, total lactase deficiency or glucose-galactose malabsorption

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Subject has to be able to produce breastmilk
Enrollment: 36 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Area under the plasma and milk concentration curve are used to calculate milk to plasma ratio | 24hours after ingestion of study drug
  M:P ratio

SECONDARY OUTCOMES:
AUC over a dosing interval | 24hours after ingestion of study drug
  AUC tau
Peak plasma concentration | Within 24 hours after ingestion of study drug
  Cmax
Concentration at the end of dosing interval | 24hours after ingestion of study drug
  Ctrough
Clearance of study drugs | 24hours after ingestion of study drug
Apparent volume of distribution | 24hours after ingestion of study drug
Half life | 24hours after ingestion of study drug

OTHER OUTCOMES:
Concentrations in breastmilk will be extrapolated to infant dosages | 24hours after ingestion of study drug

CONTACTS AND LOCATIONS:
Overall Officials: Angela Colbers, PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboudumc, Nijmegen, Netherlands